CLINICAL TRIAL: NCT00779337
Title: Epstein-Barr Virus (EBV)-Specific T Cells as Therapy for Relapsed/Refractory EBV-positive Lymphomas
Acronym: EPL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queensland Institute of Medical Research (Other)
Collaborators: The Atlantic Philanthropies (Other); Australian Department of Industry, Tourism and Resources (Industry); British Society for Haematology (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Maher Gandhi, Immunohaematology Laboratory Head, Queensland Institute of Medical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QIMR P1167; ANZCTR12608000521325
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: Epstein-Barr virus; lymphoma; immunotherapy
MeSH Terms: conditions — Lymphoma; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group study (Experimental): Autologous AdE1- Latent Membrane Protein (LMP) Cytotoxic T Lymphocytes.
  Interventions: Biological: Autologous AdE1- Latent Membrane Protein CTLs

INTERVENTIONS:
Biological: Autologous AdE1- Latent Membrane Protein CTLs — Total dose 20-800 million CTL given in 4 equal doses (5-200 million CTL) given intravenously, at weekly intervals for the first cohort of 10 patients and twice a week for the second cohort of 10 patients.

SUMMARY:
This trial will use a new method of treating lymphoma using a therapy derived from a person's Killer T cells. These Killer T cells are taken from a person's blood and grown in a test tube to increase the number of these cells that are specifically active against the lymphoma cells. The cells are then given to the patient by intravenous infusion with the aim of killing the lymphoma cells. Potentially this treatment will help to kill the residual/recurrent tumour that is present after other lymphoma treatment and reduce the chance of the tumour recurring.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* EBV-positive lymphoma as determined by in situ hybridization or equivalent (excluding Burkitts Lymphoma).
* Age 18 years or older.
* ECOG performance status 1, 2 or 3
* Life expectancy of at least 6 months.
* Measurable disease: either relapsing, partially responsive, refractory or progressive disease, includes disease detected either by clinical examination, radiographic evaluation (including CT scans, and at physician's discretion by functional imaging), or a persistently detectable plasma EBV viral load.
* No chemotherapy / radiotherapy and/or antibody therapy for at least 2 weeks prior to anticipated date of first infusion.

Exclusion Criteria:

* EBV negative tumour
* Presence of detectable malignant cells in the peripheral circulation by flow cytometry or morphology
* Serious infection within the past 28 days that has not adequately responded to therapy
* Pregnancy, or unwilling to use adequate contraception
* Serology (taken within 3 months of CTL release date) indicating active HBV or HCV infection, positive serology for HIV I&II, HTLV1 or syphilis
* Negative serology for EBV
* Psychiatric, addictive or any condition which may compromise the ability to participate in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Feasibility (generation of autologous clinical grade AdE1-LMP-specific CTL from the blood of EBV-positive lymphoma patients) | The investigational product for each participant will be assessed post production. The patient will have blood samples taken prior to and following each infusion, and then at 1, 3, 6 & 12 months following the final infusion.
Safety as assessed by adverse event monitoring. Patients will be questioned and toxicities recorded according to the International Common Toxicity Criteria. | 1 hour post 4 AdE1-LMP CTL injections (injections are weekly for first 10 participants & twice weekly for the next 10 participants), 3-5 weeks post the 4th injection, then 3, 6 and 12 months post the 4th injection
Reconstitution of EBV-specific CTL immunity with anti-viral efficacy measured by immunological & virological assessment of blood samples including immunophenotyping, intracellular cytokine assays, CD107 cytotoxicity assays and EBV DNA load analysis. | At baseline, pre and 1 hour post 4 AdE1-LMP CTL injections, 3-5 weeks post the 4th injection, then 3, 6 and 12 months post the 4th injection

SECONDARY OUTCOMES:
Optimal dose intensity of the intervention. Clinical efficacy (radiological assessment by CT), biological efficacy (reconstitution of EBV-specific CTL immunity & anti-viral efficacy), safety & efficacy of the 1st treatment schedule vs the 2nd schedule | Clinical evaluation, AE monitoring & collection of blood samples at baseline, pre & 1 hr post injections, 3-5 weeks, 3, 6 and 12 months post 4th injection. Radiological examination at baseline & at 3 to 5 wks & 3 months post the 4th treatment.
Clinical efficacy | CT scan +/- additional scans at baseline , 3-5 weeks & 3 months post the 4th injection. Clinical evaluation at baseline, pre and 1 hour post injections, 3-5 weeks, 3, 6 and 12 months post the 4th injection

CONTACTS AND LOCATIONS:
Overall Officials: Maher K Gandhi, MB CHB PhD, Principal Investigator — Queensland Institute of Medical Research
Locations (1):
- Princess Alexandra Hospital, Brisbane, Queensland, Australia